CLINICAL TRIAL: NCT04357730
Title: Fibrinolytic Therapy to Treat ARDS in the Setting of COVID-19 Infection: A Phase 2a Clinical Trial
Brief Title: Fibrinolytic Therapy to Treat ARDS in the Setting of COVID-19 Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: Genentech, Inc. (Industry); University of Colorado, Denver (Other); National Jewish Health (Other); Beth Israel Deaconess Medical Center (Other); Long Island Jewish Medical Center (Other); Scripps Health (Other); St. Mary's Medical Center (Other); University of Miami (Other); Ben Taub Hospital (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Ernest E. Moore, MD, Director of Surgical Research, Ernest E Moore Shock Trauma Center at Denver Health, Denver Health and Hospital Authority
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20-0880
Record Dates: First submitted 2020-04-18; First posted 2020-04-22 (Actual); Results first posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Severe Acute Respiratory Syndrome; Respiratory Failure; Acute Respiratory Distress Syndrome
Keywords: COVID-19; ARDS; SARS-CoV-2; Betacoronavirus
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Respiratory Insufficiency; Respiratory Distress Syndrome; COVID-19 | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Intervention Model Description: This is a Phase IIa clinical trial, open label, with a modified stepped-wedge design, testing systemic administration of fibrinolytic therapy with alteplase (tPA) versus standard of care for patients infected with COVID-19 resulting in severe respiratory failure. The design is a rapidly adaptive, pragmatic clinical trial, with 3 interim analyses and 1 final look at the data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Patients randomized to Control arm will receive no study medication; the treatment will be standard of care according to the institution's protocol for ARDS.
- Alteplase-50 bolus (Experimental): Patients randomized to Alteplase-50 group will receive 50 mg of Alteplase intravenous bolus administration over 2 hours. Re-bolusing of Alteplase, at the same dose, is permitted in those patients who show an initial transient response. The repeat dose will be given between 24 and 36 hours after the initial Alteplase administration.
  Interventions: Drug: Alteplase 50 MG [Activase]
- Alteplase-50 bolus plus drip (Experimental): Patients randomized to Alteplase-50 plus drip group will receive 50 mg of Alteplase intravenous bolus administration over 2 hours. Immediately following this initial Alteplase infusion, a drip of 2 mg/hr of Alteplase will be initiated over the ensuing 24 hours (total 48 mg infusion).
  Interventions: Drug: Alteplase 50 MG [Activase]

INTERVENTIONS:
Drug: Alteplase 50 MG [Activase] — Patients randomized to Alteplase-50 group will receive 50 mg of Alteplase intravenous bolus administration over 2 hours, given as a 10 mg push followed by the remaining 40 mgs over a total time of 2 hrs. Immediately following the Alteplase infusion, 5000 units (U) of unfractionated heparin (UFH) will be delivered and the heparin drip will be continued to maintain the activated partial thromboplastin time (aPTT) at 60-80sec (2.0 to 2.5 times the upper limit of normal). Re-bolusing of Alteplase, at the same dose, is permitted in the Alteplase-50 intervention group in those patients who show an initial transient response (>20% improvement of PaO2/FiO2 over pre-infusion of Alteplase at any of the measurements at 2, 6, 12 or 18 hours, but <50% improvement of PaO2/FiO2 at 24 hours after randomization); the repeat dose will be given between 24 and 36 hours after the initial Alteplase administration.
  Arms: Alteplase-50 bolus
Drug: Alteplase 50 MG [Activase] — wed by the remaining 40 mgs over a total time of 2 hrs. Immediately following this initial Alteplase infusion, we will initiate a drip of 2 mg/hr Alteplase over the ensuing 24 hours (total 48 mg infusion) accompanied by an infusion of 500 units per hour (U/hr) heparin during the Alteplase drip. After this, heparin dose will be increased slowly to maintain aPTT between 60 and 80 sec, titrated per attending's discretion.
  Arms: Alteplase-50 bolus plus drip

SUMMARY:
The global pandemic COVID-19 has overwhelmed the medical capacity to accommodate a large surge of patients with acute respiratory distress syndrome (ARDS). In the United States, the number of cases of COVID-19 ARDS is projected to exceed the number of available ventilators. Reports from China and Italy indicate that 22-64% of critically ill COVID-19 patients with ARDS will die. ARDS currently has no evidence-based treatments other than low tidal ventilation to limit mechanical stress on the lung and prone positioning. A new therapeutic approach capable of rapidly treating and attenuating ARDS secondary to COVID-19 is urgently needed.

The dominant pathologic feature of viral-induced ARDS is fibrin accumulation in the microvasculature and airspaces. Substantial preclinical work suggests antifibrinolytic therapy attenuates infection provoked ARDS. In 2001, a phase I trial 7 demonstrated the urokinase and streptokinase were effective in patients with terminal ARDS, markedly improving oxygen delivery and reducing an expected mortality in that specific patient cohort from 100% to 70%. A more contemporary approach to thrombolytic therapy is tissue plasminogen activator (tPA) due to its higher efficacy of clot lysis with comparable bleeding risk 8. We therefore propose a phase IIa clinical trial with two intravenous (IV) tPA treatment arms and a control arm to test the efficacy and safety of IV tPA in improving respiratory function and oxygenation, and consequently, successful extubation, duration of mechanical ventilation and survival.

DETAILED DESCRIPTION:
As the COVID-19 pandemic accelerates, cases have grown exponentially around the world. Other countries' experience suggests that 5-16% of COVID-19 in-patients will undergo prolonged intensive care with 50-70% needing mechanical ventilation(MV) threatening to overwhelm hospital capacity. ARDS has no effective treatment besides supportive care, the use of ventilation strategies encompassing low tidal volumes that limit trans-pulmonary pressures, and prone positioning in severe disease. Most current trials in clinicaltrials.gov for COVID-19-induced ARDS aim at modulating the inflammatory response or test anti-viral drugs. Sarilumab and tocilizumab that block IL-6 effects are being tested in RCT for patients hospitalized with severe COVID-19 (NCT04317092, NCT04322773, NCT04327388). The World Health Organization international trial SOLIDARITY will test remdesivir; chloroquine + hydroxychloroquine; lopinavir + ritonavir; and lopinavir + ritonavir and interferon-beta (NCT04321616). Yet studies targeting the coagulation system, which is intrinsically intertwined with the inflammatory response are lacking.

A consistent finding in ARDS is the deposition of fibrin in the airspaces and lung parenchyma, along with fibrin-platelet microthrombi in the pulmonary vasculature, which contribute to the development of progressive respiratory dysfunction and right heart failure. Similar to pathologic findings of ARDS, microthrombi have now been observed in lung specimens from patients infected with COVID-19.

Inappropriate activation of the clotting system in ARDS results from enhanced activation and propagation of clot formation as well as suppression of fibrinolysis. Our group has shown that low fibrinolysis is associated with ARDS. Studies starting decades ago have demonstrated the systemic and local effects of dysfunctional coagulation in ARDS, specifically related to fibrin. This occurs largely because of excessive amounts of tissue factor that is produced by alveolar epithelial cells and activated alveolar macrophages, and high levels of plasminogen activator inhibitor-1 (PAI-1) produced and released by endothelial cells. Consistent with this, generalized derangements of the hemostatic system with prolongation of the prothrombin time, elevated D-dimer and fibrin degradation products have been reported in severely ill COVID-19 patients, particularly in non-survivors. These laboratory findings, in combination with the large clot burden seen in the pulmonary microvasculature, mirrors what is seen in human sepsis, experimental endotoxemia, and massive tissue trauma. Targeting the coagulation and fibrinolytic systems to improve the treatment of ARDS has been proposed for at least the past two decades. In particular, the use of plasminogen activators to limit ARDS progression and reduce ARDS-induced death has received strong support from animal models, and a phase 1 human clinical trial. In 2001, Hardaway and colleagues showed that administration of either urokinase or streptokinase to patients with terminal ARDS reduced the expected mortality from 100% to 70% with no adverse bleeding events. Importantly, the majority of patients who ultimately succumbed died from renal or hepatic failure, rather than pulmonary failure.

Consideration of therapies that are widely available but not recognized for this indication and traditionally considered "high-risk" such as fibrinolytic agents is warranted in this unprecedented public health emergency, since the risk of adverse events from tPA is far outweighed by the extremely high risk of death in the patient's meeting the eligibility criteria for this trial. While the prior studies by Hardaway et al evaluating fibrinolytic therapy for treatment of ARDS used urokinase and streptokinase, the more contemporary approach to thrombolytic therapy involves the use of tissue-type plasminogen activator (tPA) due to higher efficacy of clot lysis with comparable bleeding risk to the other fibrinolytic agents.

ELIGIBILITY:
Inclusion Criteria: We will include adult patients ages 18-75 years old with known or suspected COVID-19 infection with a PaO2/FiO2 ratio < 150 or inferred PaO2/FiO2 ratio from SpO2 if ABG is unavailable (Table) persisting for > 4 hours despite optimal mechanical ventilation management according to each institution's ventilation protocols, and a neurological exam without focal signs or new deficits at time of enrollment (if patient is on paralytics, patient has been aroused sufficiently to allow a neurological examination to exclude new focal deficits or has MRI/CT scan in the last 4.5 hours with no evidence of stroke. Finally, patients must be on the ventilator for <=10 days to be eligible. Based on experience with critically ill patients, longer ventilation time may be associated with increased risk of bleeding. Patients will be enrolled based on clinical features, without consideration of language (using hospital interpreters and translated consent), race/ethnicity, or gender. A neurological exam or CT/MRI scan to demonstrate no evidence of an acute stroke is needed due to a recent case-report of large-vessel stroke as a presenting feature of COVID-19 in young individuals.

Exclusion Criteria:

* Active bleeding
* Acute myocardial infarction or history of myocardial infarction within the past 3 weeks or cardiac arrest during hospitalization
* Hemodynamic instability with Noradrenaline >0.2mcg/Kg/min
* Acute renal failure requiring dialysis
* Liver failure (escalating liver failure with total Bilirubin > 3 mg/dL)
* Suspicion of cirrhosis due to history of cirrhosis diagnosis, hepatic encephalopathy, documentation of portal hypertension, bleeding from esophageal varices, ascites, imaging or operative finding suggestive of liver cirrhosis, or constellation of abnormal laboratory test results suggestive of depressed hepatic function
* Cardiac tamponade
* Bacterial endocarditis
* Severe uncontrolled hypertension defined as SBP>185mmHg or DBP>110mmHg
* CVA (stroke), history of severe head injury within prior 3 months, or prior history of intracranial hemorrhage
* Seizure during pre-hospital course or during hospitalization for COVID-19
* Diagnosis of brain tumor, arterio-venous malformation (AVM) or ruptured aneurysm
* Currently on ECMO
* Major surgery or major trauma within the past 2 weeks
* GI or GU bleed within the past 3 weeks
* Known bleeding disorder
* P2Y12 receptor inhibitor medication (anti-platelet) within 5 days of enrollment
* Arterial puncture at a non-compressible site within the past 7 days
* Lumbar puncture within past 7 days
* Pregnancy
* INR > 1.7 (with or without concurrent use of warfarin)
* Platelet count < 100 x 109/L or history of HITT
* Fibrinogen < 300mg/dL
* Known abdominal or thoracic aneurysm
* History of CNS malignancy or CNS metastasis within past 5 years
* History of non-CNS malignancy within the past 5 years that commonly metastasizes to the brain (lung, breast, melanoma)
* Prisoner status

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2021-03-21 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ernest E Moore, MD, Principal Investigator — Denver Health Medical Center (DHMC)
Locations (9):
- United States (9):
  - Scripps Memorial Hospital La Jolla, La Jolla, California
  - University of Colorado, Denver, Aurora, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - National Jewish Health, Denver, Colorado
  - St. Mary's Medical Center, West Palm Beach, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Long Island Jewish Medical Center, New York, New York
  - Methodist Dallas Medical Center, Dallas, Texas
  - Ben Taub Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
A de-identified dataset will be made available to other investigators who may submit proposals to the PI for additional analyses or validation.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Barrett CD, Moore HB, Moore EE, Wang J, Hajizadeh N, Biffl WL, Lottenberg L, Patel PR, Truitt MS, McIntyre RC Jr, Bull TM, Ammons LA, Ghasabyan A, Chandler J, Douglas IS, Schmidt EP, Moore PK, Wright FL, Ramdeo R, Borrego R, Rueda M, Dhupa A, McCaul DS, Dandan T, Sarkar PK, Khan B, Sreevidya C, McDaniel C, Grossman Verner HM, Pearcy C, Anez-Bustillos L, Baedorf-Kassis EN, Jhunjhunwala R, Shaefi S, Capers K, Banner-Goodspeed V, Talmor DS, Sauaia A, Yaffe MB. Study of Alteplase for Respiratory Failure in SARS-CoV-2 COVID-19: A Vanguard Multicenter, Rapidly Adaptive, Pragmatic, Randomized Controlled Trial. Chest. 2022 Mar;161(3):710-727. doi: 10.1016/j.chest.2021.09.024. Epub 2021 Sep 27. PMID 34592318
- [Derived] Moore HB, Barrett CD, Moore EE, Jhunjhunwala R, McIntyre RC, Moore PK, Wang J, Hajizadeh N, Talmor DS, Sauaia A, Yaffe MB. Study of alteplase for respiratory failure in severe acute respiratory syndrome coronavirus 2/COVID-19: Study design of the phase IIa STARS trial. Res Pract Thromb Haemost. 2020 Aug 19;4(6):984-996. doi: 10.1002/rth2.12395. eCollection 2020 Aug. PMID 32838109

RESULTS

PARTICIPANT FLOW:
Period: Phase 1
Arm/Group | Control | Alteplase-50 Bolus | Alteplase-50 Bolus Plus Drip
Started | 17 | 19 | 0
Completed | 17 | 19 | 0
Not Completed | 0 | 0 | 0
Period: Phase 2
Arm/Group | Control | Alteplase-50 Bolus | Alteplase-50 Bolus Plus Drip
Started | 8 | 0 | 6
Completed | 8 | 0 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 1 Control: Phase 1 (patients 1 to 36): at randomization, patients assigned to the control group continued their current medical care according to their institution's protocols, with no input from the study team.
- Phase 1 Alteplase-50 Bolus: Phase 1 (patients 1 to 36): patients randomized to tPA-Bolus intervention received an intravenous (IV) 50mg bolus of 1mg/mL tPA as a 10mg push followed by the remaining 40mg infused over the next 2 hours. Immediately upon completion of the tPA, a 5000 unit bolus of IV unfractionated heparin (UFH) was administered and continued for the next 7 days (or until extubation) as an infusion to maintain activated partial thromboplastin time (aPTT) of 60-80 seconds. At 24 hours after tPA initiation, patients with a PaO2/FiO2 improvement that was at least 20% but did not meet the primary endpoint of a 50% improvement (i.e., 20-49% improvement) and who did not develop any of the above-mentioned exclusion criteria, received a second 50mg tPA bolus, during when the UFH infusion was halted and resumed at its prior rate as soon as the second tPA administration was complete. The heparin regimen was maintained for seven days or until successful extubation.
- Phase 2 Control: Phase 2 (patients 37 to 50): at randomization, patients assigned to the control group continued their current medical care according to their institution's protocols, with no input from the study team.
- Phase 2 Alteplase-50 Drip: Phase 2 (patients 37 to 50): patients randomized to the intervention received the tPA-Drip intervention consisting of a 50mg IV bolus of 1mg/mL tPA as a 10mg push followed by the remaining 40mg infused over the next 2 hours (not to exceed 0.9mg/kg dose). Immediately following this initial tPA infusion, patients received a drip of 2 mg/hr tPA over the ensuing 24 hours (total 48 mg infusion) accompanied by an infusion of a sub-therapeutic dose of 500U/hour of heparin during the tPA drip. Once the tPA drip terminated, the heparin dose was titrated up (no bolus) to maintain an aPTT 60-80 seconds.
- Total: Total of all reporting groups
Arm/Group | Phase 1 Control | Phase 1 Alteplase-50 Bolus | Phase 2 Control | Phase 2 Alteplase-50 Drip | Total
Number analyzed (Participants) | 17 | 19 | 8 | 6 | 50
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [57 to 62] | 59 [47 to 65] | 60.5 [51 to 65] | 64.5 [62 to 68] | 60 [52 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 2 | 0 | 13
  Male | 10 | 15 | 6 | 6 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 13 | 5 | 3 | 32
  Not Hispanic or Latino | 5 | 5 | 3 | 3 | 16
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1 | 2
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 11 | 11 | 6 | 2 | 30
  More than one race | 1 | 0 | 0 | 1 | 2
  Unknown or Not Reported | 5 | 8 | 1 | 1 | 15
BMI (body mass index) [Median (Inter-Quartile Range); unit: kg/m^2] | 36.8 [29.6 to 42] | 37.1 [32.1 to 43.7] | 30.9 [26.1 to 35.4] | 29.5 [27.7 to 36.1] | 36.8 [30.7 to 42]
Time from admission to randomization [Median (Inter-Quartile Range); unit: days] | 2 [1 to 4] | 2 [1 to 4] | 1 [0.5 to 1.5] | 5 [2 to 8] | 2 [1 to 4]
Diabetes [Count of Participants; unit: Participants] — Number of participants with diabetes mellitus
  Participants | 6 | 6 | 3 | 2 | 17
Cardiac disease [Count of Participants; unit: Participants] — Number of participants with cardiac disease
  Participants | 14 | 18 | 1 | 0 | 33
Essential hypertension [Count of Participants; unit: Participants] — Number of participants with essential hypertension
  Participants | 4 | 4 | 4 | 4 | 16
COPD [Count of Participants; unit: Participants] — Number of participants with chronic obstructive pulmonary disease (COPD)
  Participants | 13 | 15 | 0 | 3 | 31
Hyperlipidemia [Count of Participants; unit: Participants] — Number of participants with hyperlipidemia
  Participants | 6 | 5 | 1 | 1 | 13
Other comorbidities [Count of Participants; unit: Participants] — Number of participants with other comorbidities
  Participants | 5 | 7 | 5 | 4 | 21
Concurrent infections [Count of Participants; unit: Participants] — Number of participants with concurrent infections
  Participants | 10 | 13 | 5 | 4 | 32
Dexamethasone [Count of Participants; unit: Participants] — Number of participants who was treated with Dexamethasone anytime during their hospital stay.
  Participants | 11 | 9 | 3 | 3 | 26
Remdesivir [Count of Participants; unit: Participants] — Number of participants who was treated with Remdesivir anytime during their hospital stay.
  Participants | 8 | 9 | 2 | 1 | 20
Pa/FiO2 ratio [Median (Inter-Quartile Range); unit: ratio] | 107 [85 to 128.9] | 113.3 [89 to 135] | 99.5 [75.5 to 123.9] | 109.7 [77 to 132.9] | 112.3 [87 to 134.5]
National Early Warning Score (NEWS) 2 [Median (Inter-Quartile Range); unit: units on a scale] — NEWS2 is a standardised clinical scoring system developed to improve detection of deterioration in acutely ill patients. It is based on aggregate scoring of six physiological parameters; respiratory rate, oxygen saturation, systolic blood pressure, pulse rate, level of consciousness or new confusion, and body temperature. A NEWS2 score of 5 or 6 is considered a key threshold that may indicate clinical deterioration and should prompt urgent response by a clinician or a team with competence in assessment and treatment of acutely ill patients.The total score range is 0 to 20.
  units on a scale | 6 [5 to 9] | 6 [5 to 9] | 10 [7.5 to 11] | 6 [5 to 7] | 6 [5 to 9]
aPTT [Median (Inter-Quartile Range); unit: seconds] — Median activated partial thromboplastin time (aPTT)
  seconds | 30 [28.5 to 33.1] | 32.3 [26.3 to 34.9] | 31.1 [27 to 33.7] | 31 [26.7 to 41.3] | 30.5 [27.5 to 33.7]
International normalized ratio (INR) [Median (Inter-Quartile Range); unit: ratio] | 1.3 [1.1 to 1.3] | 1.1 [1.1 to 1.2] | 1.3 [1.1 to 1.3] | 1.1 [1 to 1.3] | 1.2 [1.1 to 1.3]
Fibrinogen [Median (Inter-Quartile Range); unit: mg/dL] | 668.5 [599.5 to 843] | 685 [527 to 819] | 560 [507 to 992] | 695.5 [692 to 717] | 685 [597 to 827]
D-dimer [Median (Inter-Quartile Range); unit: ng/mL] | 1900 [910 to 6137] | 2105 [1169.5 to 4294] | 4180 [1434 to 9170] | 2652 [963 to 5510] | 1900 [1089 to 4800]

OUTCOME MEASURES:

1. Primary Outcome: PaO2/FiO2 Change (Increase) From Pre-to-post Intervention
Description: PaO2/FiO2 change (increase) from pre-to-post intervention at 48 hours post randomization. Ideally, the PaO2/FiO2 will be measured with the patient in the same prone/supine position as in baseline, as change in positions may artificially reduce the change (increase) attributable to the study drug. However, given the pragmatic nature of the trial, the prone/supine position will be determined by the attending physician, in which case, we will use as an outcome the PaO2/FiO2 closest to the 48 hours obtained prior to the change in position as the outcome.
Time Frame: at 48 hours post randomization
Population: Of the 19 patients receiving the tPA-Bolus intervention, 8 required a second tPA dose due to transient PaO2/FiO2 improvement. No patients crossed over or withdrew.
Measure: Median (Inter-Quartile Range); unit: percent change
Groups:
- Phase 1 Control: At randomization, patients assigned to the control group continued their current medical care according to their institution's protocols, with no input from the study team.
- Alteplase-50 Bolus: Phase 1 (patients 1 to 36): patients randomized to tPA-Bolus intervention received an intravenous (IV) 50mg bolus of 1mg/mL tPA as a 10mg push followed by the remaining 40mg infused over the next 2 hours. Immediately upon completion of the tPA, a 5000 unit bolus of IV unfractionated heparin (UFH) was administered and continued for the next 7 days (or until extubation) as an infusion to maintain activated partial thromboplastin time (aPTT) of 60-80 seconds. At 24 hours after tPA initiation, patients with a PaO2/FiO2 improvement that was at least 20% but did not meet the primary endpoint of a 50% improvement (i.e., 20-49% improvement) and who did not develop any of the above-mentioned exclusion criteria, received a second 50mg tPA bolus, during when the UFH infusion was halted and resumed at its prior rate as soon as the second tPA administration was complete. The heparin regimen was maintained for seven days or until successful extubation.
Arm/Group | Phase 1 Control | Alteplase-50 Bolus
Number analyzed (Participants) | 17 | 19
percent change | 16.9 [-8.3 to 36.8] | 29.8 [4.5 to 88.7]

2. Primary Outcome: PaO2/FiO2 Change (Increase) From Pre-to-post Intervention
Description: as for outcome 1
Time Frame: at 48 hours post randomization
Measure: Median (Inter-Quartile Range); unit: percent change
Groups:
- Phase 2 Control: At randomization, patients assigned to the control group continued their current medical care according to their institution's protocols, with no input from the study team.
- Alteplase-50 Drip: Phase 2 (patients 37 to 50): patients randomized to the intervention received the tPA-Drip intervention consisting of a 50mg IV bolus of 1mg/mL tPA as a 10mg push followed by the remaining 40mg infused over the next 2 hours (not to exceed 0.9mg/kg dose). Immediately following this initial tPA infusion, patients received a drip of 2 mg/hr tPA over the ensuing 24 hours (total 48 mg infusion) accompanied by an infusion of a sub-therapeutic dose of 500U/hour of heparin during the tPA drip. Once the tPA drip terminated, the heparin dose was titrated up (no bolus) to maintain an aPTT 60-80 seconds.
Arm/Group | Phase 2 Control | Alteplase-50 Drip
Number analyzed (Participants) | 8 | 6
percent change | -11.9 [-24.3 to 136] | -19.6 [-21.7 to 2.3]

3. Secondary Outcome: Achievement of PaO2/FiO2 ≥ 200 or 50% Increase in PaO2/FiO2
Description: Number of Participants with Achievement of PaO2/FiO2 ≥ 200 or 50% Increase in PaO2/FiO2 (whatever is lower)
Time Frame: at 48 hours post randomization
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Control | Alteplase-50 Bolus
Number analyzed (Participants) | 17 | 19
Participants | 2 | 9

4. Secondary Outcome: Achievement of PaO2/FiO2 ≥ 200 or 50% Increase in PaO2/FiO2
Description: Number of Participants with Achievement of PaO2/FiO2 ≥ 200 or 50% Increase in PaO2/FiO2 (whatever is lower)
Time Frame: at 48 hours post randomization
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Control | Alteplase-50 Drip
Number analyzed (Participants) | 8 | 6
Participants | 3 | 1

5. Secondary Outcome: National Early Warning Score 2 (NEWS2)
Description: NEWS2 is a standardised clinical scoring system developed to improve detection of deterioration in acutely ill patients. It is based on aggregate scoring of six physiological parameters; respiratory rate, oxygen saturation, systolic blood pressure, pulse rate, level of consciousness or new confusion, and body temperature. A NEWS2 score of 5 or 6 is considered a key threshold that may indicate clinical deterioration and should prompt urgent response by a clinician or a team with competence in assessment and treatment of acutely ill patients.The total score range is 0 to 20.
Time Frame: at 48 hours post randomization
Measure: Median (Inter-Quartile Range); unit: percent change
Groups:
- Phase 1 Control: Patients randomized to Control arm will receive no study medication; the treatment will be standard of care according to the institution's protocol for ARDS.
Arm/Group | Phase 1 Control | Alteplase-50 Bolus
Number analyzed (Participants) | 17 | 19
percent change | 0 [-22.2 to 40] | 0 [-22.2 to 20]

6. Secondary Outcome: National Early Warning Score 2 (NEWS2)
Description: as for outcome 5
Time Frame: at 48 hours post randomization
Measure: Median (Inter-Quartile Range); unit: percent change
Groups:
- Phase 2 Control: Patients randomized to Control arm will receive no study medication; the treatment will be standard of care according to the institution's protocol for ARDS.
Arm/Group | Phase 2 Control | Alteplase-50 Drip
Number analyzed (Participants) | 8 | 6
percent change | -12.5 [-26.8 to 18.8] | 65.7 [0 to 80]

7. Secondary Outcome: 28 Days In-hospital Mortality
Description: 28 days mortality for hospitalized patients
Time Frame: 28 days post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Control | Alteplase-50 Bolus
Number analyzed (Participants) | 17 | 19
Participants | 5 | 4

8. Secondary Outcome: 28 Days In-hospital Mortality
Description: 28 days mortality for hospitalized patients
Time Frame: 28 days post randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Control | Alteplase-50 Drip
Number analyzed (Participants) | 8 | 6
Participants | 4 | 4

9. Secondary Outcome: ICU-free Days
Description: ICU-free days will be calculated based on (28 - number of days spent in the ICU) formula
Time Frame: 28 days of hospital stay or until hospital discharge (whichever comes first)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Phase 1 Control | Alteplase-50 Bolus
Number analyzed (Participants) | 17 | 19
days | 0 [0 to 10] | 6 [0 to 15]

10. Secondary Outcome: ICU-free Days
Description: ICU-free days will be calculated based on (28 - number of days spent in the ICU) formula
Time Frame: 28 days of hospital stay or until hospital discharge (whichever comes first)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Phase 2 Control | Alteplase-50 Drip
Number analyzed (Participants) | 8 | 6
days | 0 [0 to 0] | 0 [0 to 0]

11. Secondary Outcome: Ventilator-free Days
Description: Ventilator-free days will be calculated based on (28 - number of days on mechanical ventilation) formula.
Time Frame: 28 days of hospital stay or until hospital discharge (whichever comes first)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Phase 1 Control | Alteplase-50 Bolus
Number analyzed (Participants) | 17 | 19
days | 0 [0 to 9] | 12 [0 to 19]

12. Secondary Outcome: Ventilator-free Days
Description: Ventilator-free days will be calculated based on (28 - number of days on mechanical ventilation) formula.
Time Frame: 28 days of hospital stay or until hospital discharge (whichever comes first)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Phase 2 Control | Alteplase-50 Drip
Number analyzed (Participants) | 8 | 6
days | 0 [0 to 1] | 0 [0 to 0]

13. Post Hoc Outcome: PaO2/FiO2 Ratio at 24 Hours
Description: PaO2/FiO2 ratio measured at 24 hours post-randomization
Time Frame: 24 hours post-randomization
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Phase 1 Control | Alteplase-50 Bolus
Number analyzed (Participants) | 17 | 19
ratio | 146.7 [98.8 to 174] | 144 [122.9 to 217.1]

14. Post Hoc Outcome: PaO2/FiO2 at 24 Hours
Description: PaO2/FiO2 ratio measured at 24 hours post-randomization
Time Frame: 24 hours post-randomization
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Phase 2 Control | Alteplase-50 Drip
Number analyzed (Participants) | 8 | 6
ratio | 119.2 [111.9 to 131.3] | 94.5 [71 to 114.5]

15. Post Hoc Outcome: PaO2/FiO2 at 48 Hours
Description: PaO2/FiO2 ratio measured at 48 hours post-randomization
Time Frame: 48 hours post-randomization
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Phase 1 Control | Alteplase-50 Bolus
Number analyzed (Participants) | 17 | 19
ratio | 125 [87.5 to 147.5] | 157.1 [130 to 188]

16. Post Hoc Outcome: PaO2/FiO2 at 48 Hours
Description: PaO2/FiO2 ratio measured at 48 hours post-randomization
Time Frame: 48 hours post-randomization
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Phase 2 Control | Alteplase-50 Drip
Number analyzed (Participants) | 8 | 6
ratio | 113.7 [88.8 to 160] | 103.5 [78.8 to 105]

17. Post Hoc Outcome: aPTT at 24 Hours
Description: This outcome measure shows patients' median aPTT at 24 hours post randomization.
Time Frame: at 24 hours post randomization
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Phase 1 Control | Alteplase-50 Bolus
Number analyzed (Participants) | 17 | 19
seconds | 32.9 [28 to 36.1] | 51.7 [36.9 to 65.6]

18. Post Hoc Outcome: aPTT at 24 Hours
Description: This outcome measure shows patients' median aPTT at 24 hours post randomization.
Time Frame: at 24 hours post randomization
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Phase 2 Control | Alteplase-50 Drip
Number analyzed (Participants) | 8 | 6
seconds | 35.6 [29 to 51.2] | 27.7 [26.8 to 30]

19. Post Hoc Outcome: aPTT at 48 Hours
Description: This outcome measure shows patients' median aPTT at 48 hours post randomization.
Time Frame: at 48 hours post randomization
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Phase 1 Control | Alteplase-50 Bolus
Number analyzed (Participants) | 17 | 19
seconds | 30 [26.9 to 36.2] | 64.3 [55.7 to 73.6]

20. Post Hoc Outcome: aPTT at 48 Hours
Description: This outcome measure shows patients' median aPTT at 48 hours post randomization.
Time Frame: at 48 hours post randomization
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Phase 2 Control | Alteplase-50 Drip
Number analyzed (Participants) | 8 | 6
seconds | 53.1 [28.5 to 95.9] | 33 [28.5 to 57.4]

21. Post Hoc Outcome: Number of Patients Who Required Paralytics 48 Hours Post-randomization
Description: Number of patients who required paralytics 48 hours post-randomization
Time Frame: 48 hours post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Control | Alteplase-50 Bolus
Number analyzed (Participants) | 17 | 19
Participants | 10 | 8

22. Post Hoc Outcome: Number of Patients Who Required Paralytics 48 Hours Post-randomization
Description: Number of patients who required paralytics 48 hours post-randomization
Time Frame: 48 hours post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Control | Alteplase-50 Drip
Number analyzed (Participants) | 8 | 6
Participants | 6 | 4

23. Post Hoc Outcome: INR at 24 Hours
Description: This outcome measure shows patients' median INR at 24 hours post randomization.
Time Frame: at 24 hours post randomization
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Phase 1 Control | Alteplase-50 Bolus
Number analyzed (Participants) | 17 | 19
ratio | 1.3 [1.2 to 1.3] | 1.2 [1.1 to 1.2]

24. Post Hoc Outcome: INR at 24 Hours
Description: This outcome measure shows patients' median INR at 24 hours post randomization.
Time Frame: at 24 hours post randomization
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Phase 2 Control | Alteplase-50 Drip
Number analyzed (Participants) | 8 | 6
ratio | 1.1 [1 to 1.3] | 1.1 [1 to 1.2]

25. Post Hoc Outcome: INR at 48 Hours
Description: This outcome measure shows patients' median INR at 48 hours post randomization.
Time Frame: at 48 hours post randomization
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Phase 1 Control | Alteplase-50 Bolus
Number analyzed (Participants) | 17 | 19
ratio | 1.2 [1.1 to 1.3] | 1.2 [1.1 to 1.3]

26. Post Hoc Outcome: INR at 48 Hours
Description: This outcome measure shows patients' median INR at 48 hours post randomization.
Time Frame: at 48 hours post randomization
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Phase 2 Control | Alteplase-50 Drip
Number analyzed (Participants) | 8 | 6
ratio | 1.2 [1.1 to 1.3] | 1.2 [1.1 to 1.4]

27. Post Hoc Outcome: Fibrinogen at 24 Hours
Description: This outcome measure shows patients' median Fibrinogen (mg/dL) at 24 hours post randomization.
Time Frame: at 24 hours post randomization
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Phase 1 Control | Alteplase-50 Bolus
Number analyzed (Participants) | 17 | 19
mg/dL | 595 [521 to 828] | 627 [567 to 800]

28. Post Hoc Outcome: Fibrinogen at 24 Hours
Description: This outcome measure shows patients' median Fibrinogen (mg/dL) at 24 hours post randomization.
Time Frame: at 24 hours post randomization
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Phase 2 Control | Alteplase-50 Drip
Number analyzed (Participants) | 8 | 6
mg/dL | 588.5 [441 to 768] | 612 [542 to 822]

29. Post Hoc Outcome: Fibrinogen at 48 Hours
Description: This outcome measure shows patients' median Fibrinogen (mg/dL) at 48 hours post randomization.
Time Frame: at 48 hours post randomization
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Phase 1 Control | Alteplase-50 Bolus
Number analyzed (Participants) | 17 | 19
mg/dL | 612 [450 to 817] | 567 [520 to 786]

30. Post Hoc Outcome: Fibrinogen at 48 Hours
Description: This outcome measure shows patients' median Fibrinogen (mg/dL) at 48 hours post randomization.
Time Frame: at 48 hours post randomization
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Phase 2 Control | Alteplase-50 Drip
Number analyzed (Participants) | 8 | 6
mg/dL | 480.5 [395.5 to 638.5] | 698.5 [542 to 821]

31. Post Hoc Outcome: D-dimer at 24 Hours
Description: This outcome measure shows patients' median D-dimer (ng/mL) at 24 hours post randomization.
Time Frame: at 24 hours post randomization
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Phase 1 Control | Alteplase-50 Bolus
Number analyzed (Participants) | 17 | 19
ng/mL | 1426 [730 to 3970] | 2296 [1330 to 9700]

32. Post Hoc Outcome: D-dimer at 24 Hours
Description: This outcome measure shows patients' median D-dimer (ng/mL) at 24 hours post randomization.
Time Frame: at 24 hours post randomization
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Phase 2 Control | Alteplase-50 Drip
Number analyzed (Participants) | 8 | 6
ng/mL | 3855 [1996 to 8500] | 8477 [5540 to 11510]

33. Post Hoc Outcome: D-dimer at 48 Hours
Description: This outcome measure shows patients' median D-dimer (ng/mL) at 48 hours post randomization.
Time Frame: at 48 hours post randomization
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Phase 1 Control | Alteplase-50 Bolus
Number analyzed (Participants) | 17 | 19
ng/mL | 1326 [870 to 2970] | 1975 [1010 to 3650]

34. Post Hoc Outcome: D-dimer at 48 Hours
Description: This outcome measure shows patients' median D-dimer (ng/mL) at 48 hours post randomization.
Time Frame: at 48 hours post randomization
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Phase 2 Control | Alteplase-50 Drip
Number analyzed (Participants) | 8 | 6
ng/mL | 3480.5 [2713.5 to 4750] | 4957.5 [4261 to 7650]

35. Post Hoc Outcome: Ventilation Days
Description: Number of days patient required ventilation support
Time Frame: Duration of hospital stay, up to 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Phase 1 Control | Alteplase-50 Bolus
Number analyzed (Participants) | 17 | 19
days | 18 [9 to 28] | 13 [8 to 25]

36. Post Hoc Outcome: Ventilation Days
Description: Number of days patient required ventilation support
Time Frame: Duration of hospital stay, up to 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Phase 2 Control | Alteplase-50 Drip
Number analyzed (Participants) | 8 | 6
days | 24.5 [12 to 27] | 17.5 [16 to 25]

37. Post Hoc Outcome: Number of Participants With Adverse Events
Description: Number of Participants with Adverse Events
Time Frame: Duration of hospital stay, up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Control | Alteplase-50 Bolus
Number analyzed (Participants) | 17 | 19
Participants | 13 | 13

38. Post Hoc Outcome: Number of Participants With Adverse Events
Description: Number of Participants with Adverse Events
Time Frame: Duration of hospital stay, up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Control | Alteplase-50 Drip
Number analyzed (Participants) | 8 | 6
Participants | 5 | 2

39. Post Hoc Outcome: Number of Participants With Bleeding Events
Description: Number of Participants with Bleeding Events
Time Frame: Duration of hospital stay, up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Control | Alteplase-50 Bolus
Number analyzed (Participants) | 17 | 19
Participants | 2 | 3

40. Post Hoc Outcome: Number of Participants With Bleeding Events
Description: Number of Participants with Bleeding Events
Time Frame: Duration of hospital stay, up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Control | Alteplase-50 Drip
Number analyzed (Participants) | 8 | 6
Participants | 1 | 0

41. Post Hoc Outcome: Intensive Care Unit (ICU) Days
Time Frame: Duration of hospital stay, up to 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Phase 1 Control | Alteplase-50 Bolus
Number analyzed (Participants) | 17 | 19
days | 18 [12 to 28] | 16 [11 to 28]

42. Post Hoc Outcome: Intensive Care Unit (ICU) Days
Time Frame: Duration of hospital stay, up to 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Phase 2 Control | Alteplase-50 Drip
Number analyzed (Participants) | 8 | 6
days | 27 [12 to 30.5] | 19 [17 to 25]

ADVERSE EVENTS:
Time Frame: 28 days following randomization
Arm/Group | Control | Alteplase-50 Bolus | Alteplase-50 Drip
All-Cause Mortality (participants affected / at risk) | 11/25 | 4/19 | 5/6
Serious Adverse Events (participants affected / at risk) | 6/25 | 7/19 | 1/6
Other Adverse Events (participants affected / at risk) | 20/25 | 14/19 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=25) | Alteplase-50 Bolus (N=19) | Alteplase-50 Drip (N=6)
Arrest (Cardiac disorders) | 2 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Candidiasis (Infections and infestations) | 0 | 1 | 0
Cardiac arrhythmia (Cardiac disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Deep venous thrombosis (Vascular disorders) | 1 | 0 | 0
Failed extubation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypercalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Liver failure (Hepatobiliary disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Peritonitis (Surgical and medical procedures) | 1 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 2 | 0 | 0
Urinary track infection (Renal and urinary disorders) | 1 | 1 | 0
Worsening of lung function (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=25) | Alteplase-50 Bolus (N=19) | Alteplase-50 Drip (N=6)
ACIDOSIS (RESPIRATORY) (Metabolism and nutrition disorders) | 1 | 0 | 0
AGITATION (Nervous system disorders) | 0 | 1 | 0
ALKALOSIS METABOLIC (Metabolism and nutrition disorders) | 2 | 2 | 0
ANEMIA (Blood and lymphatic system disorders) | 5 | 4 | 0
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
BACTEREMIA (Infections and infestations) | 3 | 0 | 1
BENZODIAZEPIN/OPIATE WITHDRAWAL (Psychiatric disorders) | 0 | 1 | 0
BILIARY DILATION (Hepatobiliary disorders) | 0 | 1 | 0
BLEEDING ABDOMINAL (Gastrointestinal disorders) | 1 | 0 | 0
BLEEDING HEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
BLEEDING NASAL (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
BLEEDING ORAL (Gastrointestinal disorders) | 2 | 2 | 0
BLEEDING RECTAL TEAR (Gastrointestinal disorders) | 1 | 0 | 0
BLEEDING URINARY (Renal and urinary disorders) | 0 | 1 | 0
BLEEDING VAGINAL (Reproductive system and breast disorders) | 0 | 1 | 0
BRONCHIAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
CANDIDIASIS (Infections and infestations) | 1 | 0 | 0
CARDIAC ARRHYTMIA (Cardiac disorders) | 5 | 5 | 0
CONSTIPATION (Gastrointestinal disorders) | 2 | 5 | 0
DEHYDRATION (General disorders) | 0 | 1 | 0
DELIRIUM (Psychiatric disorders) | 6 | 3 | 0
DIARRHEA (Gastrointestinal disorders) | 2 | 2 | 0
DEEP VENOUS THROMBOSIS (Vascular disorders) | 6 | 1 | 0
DYSPHAGIA (Gastrointestinal disorders) | 0 | 2 | 0
DYSPHONIA (Ear and labyrinth disorders) | 2 | 0 | 0
EPSTEIN BARR VIRUS (Infections and infestations) | 1 | 0 | 0
ENCEPHALOPATHY (Nervous system disorders) | 2 | 0 | 0
EOSINOPHILIA (Blood and lymphatic system disorders) | 1 | 0 | 0
FACIAL EDEMA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
FAILURE TO WEAN OFF VENTILATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
FALL (General disorders) | 0 | 1 | 0
FEVER (General disorders) | 7 | 2 | 1
FRACTURE (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
HERPES SIMPLEX VIRUS (Infections and infestations) | 1 | 0 | 0
HYERPFIBRINOGENEMIA (Blood and lymphatic system disorders) | 1 | 0 | 0
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 3 | 1 | 1
HYPERKALEMIA (Metabolism and nutrition disorders) | 1 | 1 | 0
HYPERNATREMIA (Metabolism and nutrition disorders) | 2 | 3 | 0
HYPERTENSION (General disorders) | 2 | 2 | 0
HYPERVOLEMIA (General disorders) | 2 | 1 | 1
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPOKALEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPONATREMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPOTENSION (General disorders) | 9 | 4 | 0
HYPOVOLEMIA (General disorders) | 1 | 0 | 0
ILEUS (Gastrointestinal disorders) | 1 | 3 | 0
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 2 | 3 | 0
MULTIPLE ORGAN FAILURE (General disorders) | 0 | 1 | 0
MYOPATHY (Musculoskeletal and connective tissue disorders) | 6 | 5 | 0
PARAPHIMOSIS (Reproductive system and breast disorders) | 1 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
PNEUMATOCELE (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PRESSURE ULCER (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 6 | 4 | 1
RENAL TUBULAR ACIDOSIS (Renal and urinary disorders) | 1 | 0 | 0
SINUSITES (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
THROMBOCYTOSIS (Blood and lymphatic system disorders) | 0 | 2 | 0
THROMBOSIS ARTERIAL (Vascular disorders) | 1 | 0 | 0
TONGUE EDEMA (General disorders) | 0 | 0 | 1
TRANSAMINITIS (Hepatobiliary disorders) | 1 | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 1 | 2 | 0
URINARY TRACT INFECTION (Renal and urinary disorders) | 1 | 2 | 0
VOMIT (Gastrointestinal disorders) | 0 | 2 | 0
WORSENING OF LUNG FUNCTION (Respiratory, thoracic and mediastinal disorders) | 11 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/30/NCT04357730/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/30/NCT04357730/SAP_001.pdf